CLINICAL TRIAL: NCT00685594
Title: Prevention of Type 2 Diabetes With Vitamin D Supplementation in Subjects With Reduced Glucose Tolerance Detected in the Tromso Study 2007/2008
Brief Title: Vitamin D for the Prevention of Diabetes Type 2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Tromso (Other)
Collaborators: University Hospital of North Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UIT-ENDO-2008-1; NFR 184766/V50
Record Dates: First submitted 2008-05-09; First posted 2008-05-28 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Impaired Glucose Tolerance
Keywords: diabetes; vitamin D; cholecalciferol; glucose tolerance
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Cholecalciferol 20.000 IU per week for 5 years
  Interventions: Drug: cholecalciferol
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cholecalciferol — 20.000 IU cholecalciferol per week for 5 years versus placebo
  Other Names: vitamin D
  Arms: 1
Drug: Placebo — Placebo capsule once a week, identical to cholecalciferol capsule
  Arms: 2

SUMMARY:
The prevalence of type 2 diabetes is increasing, which for most societies has considerable consequences not only regarding health but also economy. Type 2 diabetes develops through a "prediabetic" stage with impaired glucose tolerance. Intervention at this stage with change in lifestyle or with medication may prevent such progression. There are indications that vitamin D is of importance in glucose metabolism, and that supplementation with vitamin D may increase both insulin secretion and insulin sensitivity. Accordingly, supplementation with vitamin D may improve glucose tolerance and potentially prevent the development of type 2 diabetes in subjects at risk. However, this has so far not been demonstrated in a prospective, randomised clinical study. In the present study we will therefore include 600 subjects with impaired glucose tolerance (or impaired fasting glucose) detected in the Tromso study 2007/2008 and randomize to supplementation with vitamin D 20.000IU per week or placebo for 5 years. A glucose tolerance test will be performed each year, and development of type 2 diabetes will be the main endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance

Exclusion Criteria:

* Serious heart disease
* Renal stone disease
* Hypercalcemia
* Sarcoidosis

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2008-03; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
development of diabetes type 2 | 5 years

SECONDARY OUTCOMES:
change in glucose metabolism | 5 years
change in lipid status | 5 years
change in mood | 5 years
change in BMD hip | 5 years
change in intima media thickness carotid artery | 5 years
change in frequency of infections | 5 years
change in blood pressure | 5 years
Change in Insulin sensitivity | 5 years
change in HbA1c | 5 years
change in weight | 5 years
change in telomer length | 5 years

OTHER OUTCOMES:
Oral glucose tolerance response to vitamin D supplementation in relation to polymorphisms in the vitamin D system | 1 year
  The response to oral glucose tolerance test (fasting and 2 h blood glucose, serum insulin, C-peptide, measures of insulin resistiance as well as metabolic parameters (lipids, blood pressure)) will be evaluated in the results at the 1-year visit in relation to genetic polymorphisms in the vitamin D system

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- University of Tromso, Tromsø, Norway

REFERENCES:
- [Derived] Jorde R, Sollid ST, Svartberg J, Schirmer H, Joakimsen RM, Njolstad I, Fuskevag OM, Figenschau Y, Hutchinson MY. Vitamin D 20,000 IU per Week for Five Years Does Not Prevent Progression From Prediabetes to Diabetes. J Clin Endocrinol Metab. 2016 Apr;101(4):1647-55. doi: 10.1210/jc.2015-4013. Epub 2016 Feb 1. PMID 26829443